CLINICAL TRIAL: NCT01261403
Title: A Phase 2, Randomized, Double- Blind, Placebo-controlled, Multi-center Study to Evaluate the Safety and Efficacy of Intravenous Infusion of Human Placenta-Derived Cells (PDA001) for the Treatment of Adults With Active Rheumatoid Arthritis
Brief Title: Study of Human Placenta-derived Cells (PDA001) to Evaluate the Safety and Effectiveness for Patients With Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment terminated pending additional Phase 1 data
Sponsor: Celularity Incorporated (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCT-PDA001-RA-001
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Human Placenta-Derived Cells
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): 1 Unit of PDA001 or 4 units Vehicle Control intravenous on Day 0 and Day 7
  Interventions: Biological: PDA001; Drug: Vehicle Controlled Placebo
- Group 2 (Experimental): 4 Units PDA001 or 4 units Vehicle Control intravenous (Placebo) on Day 0 and Day 7
  Interventions: Biological: PDA001; Drug: Vehicle Controlled Placebo
- Vehicle control (Placebo Comparator): Placebo - Vehicle Control Arm
  Interventions: Drug: Vehicle Controlled Placebo

INTERVENTIONS:
Biological: PDA001 — Dose escalation study: Subjects will be assigned to 1 of 2 treatment groups (1 unit or 4 units vs. vehicle control) based on the order in which they enroll in the study. Intravenous infusion will be administered on days 0 and 7. Nonresponders will be unblinded after 12 weeks of study. Non- responders on vehicle control will be re-dosed with the active PDA001 dose assigned at baseline (2 infusions, 7 days apart). Nonresponders taking active PDA001 will enter the safety follow-up portion of the study. Responders at 12 weeks will continue in the safety and efficacy follow-up portion of the study until 12 months of study. Responders will be treated for RA flare between 3-9 months of study with the active PDA001 dose assigned at baseline (2 infusions, 7 days apart).
  Arms: Group 1; Group 2
Drug: Vehicle Controlled Placebo — Cohort Dose Level 1: 4 units vehicle controlled placebp infused on Day 0 and Day 7
  Cohort Dose Level 2: 4 units vehicle controlled placebo infused on Day 0 and Day 7

SUMMARY:
The primary objective of the study is to assess the safety and efficacy of 2 dose groups (PDA001 versus vehicle control) in subjects with active rheumatoid Arthritis. The secondary objectives of the study are to determine the clinical response at defined visit intervals, determine the time to flare of RA symptoms and to quantify changes in inflammatory markers including C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), serum amyloid A (SAA), and IL-6.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Diagnosis of RA as defined by the 1987-revised ACR criteria.
2. RA, characterized by at least 6 out of 66 swollen joints and 6 out of 68 tender joints at Screening and Baseline, and at least 2 of the following: a C reactive protein level (CRP), greater than the upper limit of normal (ULN) ³ 1 mg/dl, an erythrocyte sedimentation rate (ESR) of at least 28 mm per hour, or morning stiffness lasting longer than 45 minutes.
3. Non responsive or intolerant to a minimum of 2 RA therapies which are classified as DMARDs, biologics, or corticosteroids.
4. Biological medication must be discontinued 30 day prior to the first dose of study drug, except golimumab and actemra which are 60 days, and infliximab, alefacept and efalizumab, which must have been discontinued 90 days prior to the first dose of IP.
5. Cytotoxic agents, including but not limited to chlorambucil, cyclophosphamide, nitrogen mustard, or other alkylating agents must have been discontinued 90 days prior to the first dose of IP.
6. Subjects must be able to tolerate intravenous infusions in both arms.
7. There should be no change in RA medication dose anticipated during the initial treatment and re treatment periods and the respective 12 week follow-up period for each dosing treatment period. The following rules apply for anti-rheumatic medications taken during the study:
8. DMARDs must have must have been stable for least 90 days prior to dosing with IP.
9. Low -dose corticosteroids are permitted (prednisolone ≤ 10 mg per day or equivalent). Corticosteroids must have been stable for at least 30 days prior to dosing with IP.
10. DMARDs and corticosteroids must remain stable throughout the initial 3 months of study and throughout subsequent treatment periods

The presence of any of the following will exclude a subject from enrollment:

1. Prior use of rituximab and other B-cell depleting therapies, abatacept, prior use of more than 2 biologic therapies.
2. Subject has received an investigational agent in any indication-within 60 days (or 5 half-lives, whichever is longer) prior to treatment with IP.
3. Subject has received previous cell therapy.
4. Serum creatinine concentration > 2.0 mg/dl at screening.
5. Alkaline phosphatase > 2.5x the upper limit of normal at screening.
6. Bilirubin level > 1.5 mg/dL (unless subject has known Gilbert's disease).
7. Untreated chronic infection or treatment of any infection with antibiotics within 4 weeks prior to dosing with IP.
8. Positive HIV test at Screening. Positive Hepatitis B surface antigen at Screening. Positive Hepatitis C antibody at Screening.
9. Organic heart disease (e.g., congestive heart failure), myocardial infarction within six (6) months prior to screening or clinically significant findings on ECG at screening. Clinically significant arrhythmia.
10. Primary or secondary immunodeficiency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number/Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response within 12 weeks following the initial dose of study drug | Baseline through Week 12
  A participant is a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in 68 tender joint count; • ≥ 20% improvement in 66 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: o Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]) o Patient's global assessment of disease activity (measured on a 100 mm VAS) o Physician's global assessment of disease activity (measured on a 100 mm VAS) o Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)) o C-Reactive Protein

SECONDARY OUTCOMES:
Number/Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at 6 months | Baseline and 6 months
  A participant is a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in 68 tender joint count; • ≥ 20% improvement in 66 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: o Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]) o Patient's global assessment of disease activity (measured on a 100 mm VAS) o Physician's global assessment of disease activity (measured on a 100 mm VAS) o Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)) o C-Reactive Protein
Number/percent of subjects achieving an ACR 20 clinical response at each scheduled visit during the first 12 months following the first infusion of study drug. | Baseline and each scheduled visit through 12 months following the first infusion of study drug
  A participant is an ACR 20 responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in 68 tender joint count; • ≥ 20% improvement in 66 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: o Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]) o Patient's global assessment of disease activity (measured on a 100 mm VAS) o Physician's global assessment of disease activity (measured on a 100 mm VAS) o Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)) o C-Reactive Protein
Number/percent of subjects achieving an ACR 50 clinical response at each scheduled visit during the first 12 months following the first infusion of study drug. | Baseline and each scheduled visit through 12 months following the first infusion of study drug.
  A participant is an ACR responder if the following 3 criteria for improvement from Baseline were met: • ≥ 50% improvement in 68 tender joint count; • ≥ 50% improvement in 66 swollen joint count; and • ≥ 50% improvement in at least 3 of the 5 following parameters: o Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]) o Patient's global assessment of disease activity (measured on a 100 mm VAS) o Physician's global assessment of disease activity (measured on a 100 mm VAS) o Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)) o C-Reactive Protein
Number/percent of subjects achieving an ACR 70 clinical response at each scheduled visit during the first 12 months following the first infusion of study drug. | Baseline and each scheduled visit through 12 months following the first infusion of study drug.
  A participant is an ACR 70 responder if the following 3 criteria for improvement from Baseline were met: • ≥ 70% improvement in 68 tender joint count; • ≥ 70% improvement in 66 swollen joint count; and • ≥ 70% improvement in at least 3 of the 5 following parameters: o Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]) o Patient's global assessment of disease activity (measured on a 100 mm VAS) o Physician's global assessment of disease activity (measured on a 100 mm VAS) o Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)) o C-Reactive Protein
Number/percent of subjects achieving a clinical response based on their Clinical Disease Activity Index (CDAI) at each scheduled visit during the first 12 months following the first infusion of study drug. | Baseline and each scheduled visit through 12 months following the first infusion of study drug
  A subject is considered a responder based on the Clinical Disease Activity Index (CDAI): A composite index where CDAI = SJC+TJC+SGA+PGA. SJC and TJC are the numbers of swollen and tender joints based on 28-joint counts; SGA and PGA represent the subject's and physician's global assessment of disease activity. The CDAI score ranges from 0-76. Clinical disease activity is defined according to CDAI scores where Remission is ≤ 2.8, Low Disease Activity > 2.8 and ≤ 10, Moderate Disease Activity > 10 and ≤ 22, and High Disease Activity > 22
Number/percent of subjects achieving a clinical response based on their Disease Activity Score (DAS 28) score at each scheduled visit during the first 12 months following the first infusion of study drug | Baseline and each scheduled visit through 12 months following the first infusion of study drug
  A subject is considered a responder based on Disease Activity Score 28 (DAS 28): A measure of severity of disease derived from the following: 28 tender joint count (TJC28); 28 swollen joint count (SJC28), which do not include the distal interphalangeal (DIP) joints, the hip joint, or the joints below the knee, CRP, and SGA. A DAS 28 score > 5.1 indicates high disease activity, a DAS28 score < 3.2 indicates low disease activity, and a DAS28 score < 2.6 indicates clinical remission
Number/Percent of Participants Who Achieve the European League Against Rheumatism (EULAR) Response Criteria Using CRP at Month 12 | Baseline and each scheduled visit through 12 months following the first infusion of study drug.
  A subject is considered a responder based on EULAR response: The EULAR response criteria classify each subject as a good, moderate or non-responder to treatment based on the degree of improvement from baseline and the level of disease activity at the endpoint. EULAR response is derived using the individual subject's DAS28 as the measure of severity of disease. Good or moderate response is defined as follows: Good response: DAS28 at the time point ≤ 3.2 and improvement from baseline > 1.2 Moderate response: DAS28 at the time point > 3.2 and improvement from baseline > 1.2, or DAS28 at the time point ≤ 5.1 and improvement from baseline > 0.6 and ≤ 1.2
The change from baseline in the ACR core components. ACR Core Component #1: Percentage Change From Baseline in the Swollen Joint Count at each scheduled visit. | Baseline and each scheduled visit through 12 months following the first infusion of study drug
  Joint tenderness is the presence of pain in a joint when pressure is applied by the examiner to elicit tenderness. The 68 tender joint count evaluates the following joints: upper-temporomandibular, sternoclavicular, acromioclavicular, shoulder, elbow, wrist, meta-carpophalangeal, proximal interphalangeal and distal interphalangeal; lower: hip, knee, ankle, midtarsal, metatarsophalangeal and proximal interphalangeal.
ACR Core Component #2: Percentage Change From Baseline in the Swollen Joint Count at each scheduled visit through Month 12 following the initial infusion of study drug | Baseline and at each scheduled visit through Month 12 following the initial infusion of study drug
  Joint swelling is soft tissue swelling that is detectable along the joint margins and is assessed by inspection and direct palpation of the joint, by the examiner. The ACR 66 swollen joint count evaluates the following joints: upper-temporomandibular, sternoclavicular, acromioclavicular, shoulder, elbow, wrist, metacarpophalangeal, proximal interphalangeal and distal interphalangeal; lower: knee, ankle, midtarsal, metatarsophalangeal and proximal interphalangeal.
ACR Core Component #3 Percentage Change From Baseline in the Subject Assessment of Pain at each scheduled visit through Month 12 following the initial dose of study drug | Baseline and at each scheduled visit through Month 12 following the initial dose of study drug
  The Subject Assessment of Pain was measured asking the participant to place a vertical line on a 100-mm visual analog scale on which the left-hand boundary (score = 0 mm) represents "no pain," and the right-hand boundary (score = 100 mm) represents "pain as severe as can be imagined." The distance from the mark to the left-hand boundary was recorded in millimeters.
ACR component #4 Percentage Change From Baseline in the Subject Global Assessment of Disease Activity at each scheduled visit through Month 12 following the initial dose of study drug | Baseline and at each scheduled visit through Month 12 following the initial dose of study drug
  The Subject Global Assessment of Disease Activity was measured asking the participant to place a vertical line on a 100-mm visual analog scale on which the left-hand boundary (score = 0 mm) represents " lowest disease activity," and the right-hand boundary (score = 100 mm) represents " highest disease activity." The distance from the mark to the left-hand boundary was recorded in millimeters.
ACR Component #5 Percentage Change From Baseline in the Physician Global Assessment of Disease Activity at each scheduled visit through Month 12 following the initial dose of study drug | Baseline and Month 12
  The Physician Global Assessment of Disease Activity was measured asking the physician to assess the subject's current arthritis disease activity by placing a vertical line on a 100-mm visual analog scale on which the left-hand boundary (score = 0 mm) represents " lowest disease activity," and the right-hand boundary (score = 100 mm) represents " highest disease activity." The distance from the mark to the left-hand boundary was recorded in millimeters
ACR Component #6; Percentage Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at each scheduled visit through Month 12 following the initial dose of study drug | Baseline and at each scheduled visit through Month 12 following the initial dose of study drug
  The Health Assessment Questionnaire - Disability Index (HAQ-DI) was a patient-reported questionnaire consisting of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from baseline in the overall score indicate improvement in functional ability.
ACR Component#7 Percentage Change From Baseline in the High Sensitivity C-Reactive Protein (CRP) at each scheduled visit through Month 12 following the initial dose of study drug | Baseline at each scheduled visit through Month 12 following the initial dose of study drug
  C-Reactive Protein (CRP) is a substance produced by the liver that increases in the presence of inflammation in the body. An elevated CRP level is identified with blood tests and is considered a non-specific "marker" for disease
ACR Component #8 Percentage Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at each scheduled visit through Month 12 following the initial dose of study drug | Baseline and at each scheduled visit through Month 12 following the initial dose of study drug
  The erythrocyte sedimentation rate (ESR) is a blood test that can reveal inflammatory activity. The subject's blood is placed in a tall, thin tube, red erythrocytes gradually settle to the bottom. Inflammation can cause the cells to clump together. Because these clumps of cells are denser than individual cells, they settle to the bottom more quickly. The ESR test measures the distance red blood cells fall in a test tube in one hour. The farther the red blood cells have descended, the greater the inflammatory response
Change from baseline in rheumatoid factors at each scheduled visit through Month 12 following the initial dose of study drug | Baseline and each scheduled visit through Month 12 following the initial dose of study drug
  Rheumatoid factor is an antibody that is measurable in the blood. Rheumatoid factor is actually an antibody that can bind to other antibodies. High levels of rheumatoid factor can indicate a tendency toward more aggressive disease and/or a tendency to develop rheumatoid nodules and rheumatoid lung disease.
Time to flare of Rheumatoid Arthritis (RA) symptoms | At defined intervals
  A flare is defined as a 20% increase in both tender and swollen joint counts, an increase in Physician Global Assessment of Disease ≥ 20 mm and an increase in at least 1 of 2 criteria (Patient Global Assessment of Disease ≥ 20 mm, Patient Assessment of Pain ≥ 20 mm) when compared with corresponding values from the subject's best response. Best response is determined by the subject's lowest CDAI score
Changes in inflammatory markers including C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), serum amyloid A (SAA), and IL-6 | At defined intervals
  Inflammatory markers are certain laboratory tests performed using the subjects' serum that indicate the presence of RA. Changes in these test results may indicate an improvement in RA
Change From Baseline in the Disease Activity Score 28 (DAS 28) Using CRP | Baseline and Month 6
  The DAS28 measures the severity of disease at a specific time and is derived from the following variables: • 28 tender joint count (TJC28) • 28 swollen joint count (SJC28), which do not include the distal interphalangeal (DIP) joints, the hip joint, or the joints below the knee; • C-reactive protein (CRP) • Subject's global assessment of disease activity (SGA). A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission. Remission: ≤ 2.8; Low Disease Activity: > 2.8 and ≤ 10; Moderate Disease Activity: > 10 and ≤ 22; High Disease Activity: > 22
Change From Baseline in the Clinical Disease Activity Index (CDAI) at Month 3 | Baseline and Month 3
  Clinical Disease Activity Index (CDAI): A simplified composite index as defined by: CDAI = SJC + TJC + SGA + PGA) • SJC and TJC are the numbers of swollen and tender joints based on 28-joint counts. • SGA and PGA represent the subject's and physician's global assessment of disease activity. o The CDAI score ranges from 0-76. Clinical disease activity is categorized according to CDAI scores where Remission ≤ 2.8, Low Disease Activity > 2.8 and ≤ 10, Moderate Disease Activity > 10 and ≤ 22, and High Disease Activity > 22
Change From Baseline in the Clinical Disease Activity Index (CDAI) at Month 6 | Baseline and Month 6
  Clinical Disease Activity Index (CDAI): A simplified composite index as defined by: CDAI = SJC + TJC + SGA + PGA) • SJC and TJC are the numbers of swollen and tender joints based on 28-joint counts. • SGA and PGA represent the subject's and physician's global assessment of disease activity. o The CDAI score ranges from 0-76. Clinical disease activity is categorized according to CDAI scores where Remission ≤ 2.8, Low Disease Activity > 2.8 and ≤ 10, Moderate Disease Activity > 10 and ≤ 22, and High Disease Activity > 22

CONTACTS AND LOCATIONS:
Overall Officials: Solveig Ericson, MD, Study Director — Celularity Incorporated
Locations (16):
- United States (16):
  - Pinnacle Research Group, Anniston, Alabama
  - Advanced Pain Research Institute, Arcadia, California
  - UCLA, Los Angeles, California
  - Desert Medical Advances, Palm Desert, California
  - Sanitas Research, Coral Gables, Florida
  - Compass Research, LLC, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Four Rivers Clinical Research Inc., Paducah, Kentucky
  - Arthritis and Diabetes Clinic, Inc, Monroe, Louisiana
  - St. Paul Rheumatology, PA, Eagan, Minnesota
  - SNS Rheumatology, Lakewood, New Jersey
  - David R. Mandel, MD, Inc., Mayfield, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Health Research Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas